CLINICAL TRIAL: NCT04112355
Title: Establishing the Dynamic Range of Healthy Pediatric Inflammatory Responses to Vaccinations and Identifying the Role of IL1RN Polymorphisms in Controlling This Response.
Brief Title: Measuring the Healthy Pediatric Inflammatory Response to Vaccination.
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles L. Howe, Principal Investigator, Mayo Clinic
Other Study IDs: 19-001219
Record Dates: First submitted 2019-04-08; First posted 2019-10-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for this study. Tests done only for research purposes are not meant to provide clinical information or help care for participants. The results are only important for research. Therefore, the results of tests will not be provided to participants. In the rare event that a finding might affect the health of a participant, the investigators will offer additional information. If the participant decides to follow up and further medical testing or care is needed, the costs will be the responsibility of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6 months of age: Visit 1
  This visit will take about 15 minutes and will be at the time of the next scheduled clinical vaccinations. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Provided a temperature diary to fill out for the next week Visit 2
  This visit will take about 15 minutes and will be approximately 7 days after the first visit. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Collect temperature diary if not already mailed in
  Interventions: Other: Blood Collection
- 12 months of age: Visit 1
  This visit will take about 15 minutes and will be at the time of the next scheduled clinical vaccinations. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Provide a temperature diary to fill out for the next week Visit 2
  This visit will take about 15 minutes and will be approximately 7 days after the first visit. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Collect temperature diary if not already mailed in
  Interventions: Other: Blood Collection
- 5 years of age: Visit 1
  This visit will take about 15 minutes and will be at the time of the next scheduled clinical vaccinations. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Provide a temperature diary to fill out for the next week Visit 2
  This visit will take about 15 minutes and will be approximately 7 days after the first visit. Study procedures at this visit include :
  * Draw a blood sample based on age groups below
  * Collect temperature diary if not already mailed in
  Interventions: Other: Blood Collection

INTERVENTIONS:
Other: Blood Collection — Blood draw

SUMMARY:
The purpose of this research is to understand the normal healthy response to immunological challenge by measuring circulating cytokine and chemokine levels before and after vaccinations in healthy children. These data will define a range of normal responses that can be used to help us understand pathogenic mechanisms in children who do not respond normally to infections. In addition, this study will test the hypothesis that genetic polymorphisms in the interleukin-1 receptor antagonist gene are associated with differential inflammatory responses across the healthy spectrum.

DETAILED DESCRIPTION:
Children who experience seizures that cannot be stopped by traditional anti-seizure medications often suffer profound brain injury and intellectual disability. Indeed, many of these children do not survive. In one study, 12% of children who developed an acute onset disease called FIRES (febrile infection-related epilepsy syndrome) died during the early stages of the disease, and of the children who survived, more than 90% developed cognitive impairment and lifelong epilepsy that could not be treated by our standard drugs. The discovery of new therapeutic strategies is therefore imperative.

A role for inflammation and the innate and adaptive immune systems in generating seizures is a burgeoning but understudied field in epilepsy research. While data from multiple human and animal studies suggests that inflammatory cytokines can drive ictogenesis, the development of strategies to modulate inflammation are hindered by insufficient knowledge regarding the dynamic range of healthy responses to infection and immunological challenge. On this basis, the investigators intend to measure changes in levels of inflammatory cytokines and chemokines in the blood induced by the normal healthy response to vaccination. To do so, the investigators will collect a small amount of blood from children just before they receive their standard vaccinations at 6 months, 12 months, or 4-6 years of age. A follow-up sample will then be collected from the same children approximately 10-14 days later. Since it is known that about 30% of children develop a fever within this timeframe, it is expected that the size of the change in inflammatory factors in each child will reflect a Gaussian distribution, with "high responders" and "low responders" centered on a mean response. For each sample the investigators will isolate serum and measure the levels of interleukin-1 beta, interleukin-6, tumor necrosis factor alpha, chemokine (C-C motif) ligand 2, chemokine (C-C motif) ligand 5, chemokine (C-X-C motif) ligand 1, chemokine (C-X-C motif) ligand 2, chemokine (C-X-C motif) ligand 8, chemokine (C-X-C motif) ligand 9, and chemokine (C-X-C motif) ligand 10.

In addition, based on recent findings showing that some children with acute seizure disorders exhibit previously unknown genetic polymorphisms in the interleukin-1 receptor antagonist (IL1RA) gene that are associated with altered immunological function, the investigators have hypothesized that normal healthy children will exhibit a spectrum of IL1RA function that will correlate with the size of their response to vaccination. To test this hypothesis the investigators will collect genomic DNA for sequencing of the IL1RA gene (also known as IL1RN) and will measure the function of the IL1RA protein in serum. This genetic and functional data will be correlated with the inflammatory cytokine and chemokine response measured in serum.

Several key findings will be made in this study.

1. Measure the normal range of inflammatory responses that occur in the blood when a person is given a vaccine; blood will be collected just before the vaccination and then again 1-2 weeks later.
2. Measure protein function in the blood and build up a graph showing the range of such function in healthy kids.
3. Sequence the gene that produces a specific protein in healthy children. All humans have minor changes in genes that subtly alter the function of proteins. These are called polymorphisms and they are completely normal. The investigators want to build up a picture of the type of polymorphisms that occur in children and then compare these differences. This information might help to someday develop new ways to help children with dysfunctional proteins.

This study is in no way based on the idea that vaccines "are bad". This study was designed because children all respond a little differently to vaccines (for example, some get sore at the injection site, some get a low fever, some feel more tired than usual) and this indicates that the body is responding to the immunization in ways that can be measured. The investigators think that the normal healthy response to vaccination will help define a range of responses that can be used to help other children who do not respond normally to infections. While this study is focused on a specific protein and on helping children who have defects in this factor, these findings will be widely relevant to understanding many diseases of the immune system in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-7 months of age receiving the 3rd scheduled dose of the diphtheria, tetanus, pertussis, inactivated polio, Haemophilus influenzae type b, and pneumococcal conjugate vaccine (DTap-IPV/Hib+PCV13).
* Children 10-18 months of age receiving the 1st scheduled dose of the measles, mumps, rubella, and varicella vaccine (MMR+VZV).
* Children 4-6 years of age receiving the 2nd scheduled MMR+VZV dose.
* Children and young adults receiving the annual flu vaccine or COVID vaccine

Exclusion Criteria:

* History of autoinflammatory or autoimmune disease.
* History of genetic or metabolic disorder.
* History of hematological disorder.
* History of malignancy or active malignancy undergoing suppressive treatment.
* Blood donation or collection within 8 weeks of the study.
* Signs or symptoms consistent with severe infection at the time of first visit.
* Weight less than 6 kg in group 1, less than 7.5 kg for group 2, less than 12 kg for group 3.

Ages: 4 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children scheduled for vaccinations at Mayo Clinic in Rochester, MN
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes in normal pediatric interleukin-1 beta levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum interleukin-1 beta levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric interleukin-6 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum interleukin-6 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric tumor necrosis factor-alpha levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum tumor necrosis factor-alpha levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-C motif) ligand 2 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-C motif) ligand 2 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-C motif) ligand 5 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-C motif) ligand 5 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-X-C motif) ligand 1 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-X-C motif) ligand 1 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-X-C motif) ligand 2 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-X-C motif) ligand 2 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-X-C motif) ligand 8 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-X-C motif) ligand 8 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-X-C motif) ligand 9 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-X-C motif) ligand 9 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Changes in normal pediatric chemokine (C-X-C motif) ligand 10 levels in serum at 1 week after immunization relative to baseline. | Baseline, 1week
  Measurement of serum chemokine (C-X-C motif) ligand 10 levels will be analyzed and compared between the pre-immunization and post-immunization timepoints. Response profiles will also be compared between subjects.
Determine the range of normal single nucleotide polymorphisms in the interleukin-1 receptor antagonist (IL-1RN) gene. | Baseline
  The IL-1RN gene will be sequenced from genomic DNA. Sequences will be compared between subjects and associated with cytokine and chemokine levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No